CLINICAL TRIAL: NCT07114744
Title: Early Cochlear Implant Use
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-01603; K99DC021727 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Implant Users

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly Implanted Users: Participants have no prior experience with cochlear implants (recruitment happens prior to cochlear implantation) will complete at home testing (~25 sessions) over ~3 months of implant use.
  Interventions: Other: Take home tests
- Experienced Cochlear Implant Users: Participants who have used the same stimulation strategy since initial stimulation will complete at home testing (~25 sessions) over ~3 months of implant use.
  Interventions: Other: Take home tests

INTERVENTIONS:
Other: Take home tests — These tests will test the discriminability of sounds that vary systematically along the frequency and temporal dimensions of sound. Over the course of the 3 months post-activation, subjects will self-complete "take-home" tests at location of their choosing. Each test session will include the entire test-battery will be repeated frequency as often as every day and then reducing frequency of testing corresponding to the rate of speech perception improvement.

SUMMARY:
This observational study will examine newly activated cochlear implant users and determine whether their abilities to discern simple sounds change and relate to improved speech perception. Take-home computers and test-equipment will be sent home, and subjects will complete approximately 25 test sessions over the first 3 months of cochlea implant use. Then, subjects will be tested 3 more times in the laboratory until 1 year-post activation. The primary objective is to determine and quantify how sounds change and speech perception improves over the course of early cochlear implant use.

ELIGIBILITY:
Inclusion Criteria:

1. Postlingually deaf cochlear implant users
2. severe or profound hearing loss
3. who do not have other diagnoses communicative or cognitive disorders.
4. Test population: no prior experience with cochlear implants (recruitment happens prior to cochlear implantation).
5. Control population: subjects who have used the same stimulation strategy since initial stimulation, who note no continuing improvements or changes with their devices with respect to speech comprehension.

Exclusion Criteria:

1. Diagnosed cognitive or communicative disorders (other than deafness)
2. Below 18 years of age
3. Above the age of 85 years old.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes hearing impaired adults. Both genders will be recruited. All subjects will be recruited from the NYU Cochlear Implant Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of correct responses during speech perception tests | Baseline, 1 year
  Speech perception tests involves presentation of a speech stimulus (may be a word, sentence, nonsense words, or other speech sounds) and subjects will have to indicate what they heard. The total score is the percentage of speech stimulus correctly understood, ranging from 0-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A. Svirsky, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to:ariel.hight@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to ariel.hight@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.